CLINICAL TRIAL: NCT06882018
Title: Educational Strategies for Maintaining Technical Skills in Neonatal Resuscitation for the Nursing Team: A Pilot Project
Brief Title: Educational Strategies for Maintaining Technical Skills in Neonatal Resuscitation for the Nursing Team
Acronym: Neo-VPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Moussa (Other)
Responsible Party: Sponsor-Investigator, Ahmed Moussa, Neonatalogist, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-7607
Record Dates: First submitted 2024-12-19; First posted 2025-03-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ventilation Therapy; Complications; Technical Skills; Nurse's Role

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated practice guided by peers (Experimental): Intervention group which will use the educational tool during repeated practice guided by peers
  Interventions: Other: Repeated practice guided by peers
- Instructor-guided deliberate practice (Active Comparator): A control group that will use the traditional method, instructor-guided deliberate practice
  Interventions: Other: Instructor-guided deliberate practice

INTERVENTIONS:
Other: Repeated practice guided by peers — This approach involves repeated, peer-guided practice. Each session will involve two participants, who will support each other using the feedback grid from the first section of the "Neonatal Mask Ventilation Competency Assessment Tool" developed by DiLabio et al. (2018) to provide feedback on practicing technical skills.
  Arms: Repeated practice guided by peers
Other: Instructor-guided deliberate practice — In this group, practice is deliberate (PD) and is led by an instructor. Each session will be supervised by an instructor for two to four participants, and the latter will use the same feedback grid as that used in the intervention group to provide feedback.
  Arms: Instructor-guided deliberate practice

SUMMARY:
Despite efforts for initial training in neonatal resuscitation, health professionals show a decline in post-training skills, requiring continuing training. This randomized controlled pilot study will compare the feasibility and preliminary effects of two educational tools in the field, namely the traditional teaching method (instructor-assisted deliberate practice) and an educational tool developed during the research project that involves repeated peer-guided practice. Both groups will perform the same educational activity using a mobile training station equipped with the equipment necessary for the PPV. Each session will be of 30 minutes and will be repeated three times over a period of three months.

DETAILED DESCRIPTION:
Background :

Despite efforts for initial training in neonatal resuscitation (NR), health professionals show a decline in post-training skills, requiring continuing training. Lack of practice, financial resources and competent worker are the main challenges encountered on the department. However, optimal care in NR, particularly in positive pressure ventilation (PPV) saves lives. Deliberate practice (DP) is a simulation-based instructional strategy known for its effectiveness in maintaining skills. However, DP is limited by the resources and costs linked to the presence of experts. Self-directed, learner-centred approaches could solve these challenges.

This pilot study seeks to compare the proposed tool with a traditional method which is learning through PD guided by an instructor. This feasibility study will make it possible in the future to plan more in-depth research to promote the possibility of generalization.

Th specific research objectives are as follows.

* The primary objective is to document the feasibility of implementing the proposed educational tool in order to maintain technical skills in VPP among practising nurses by comparing it to the traditional method. Feasibility measures include participant satisfaction with the quality of the teaching method, speed of participant recruitment, and participant participation and retention rate.
* The secondary objective is to evaluate whether the participants' confidence in VPP, the propensity to change one's own practice as well as the performance of VPP in the experimental group is similar to the traditional group.

Methods

* Design This randomized controlled pilot study will compare the feasibility and preliminary effects of two educational tools.
* Sample and setting The research project will take place in the neonatal intensive care unit of the Sainte-Justine Hospital Centre (CHUSJ). The target population is the nursing team which includes approximately 240 people. The level of expertise of the sample aims to be as variable as the current population of the neonatal intensive care nursing team.

Convenience sampling due to its pragmatic approach. It allows to recruit accessible participants on time and with limited resources. A stratified randomization will be used to optimize the balance of the groups taking into account the two types of professionals (registered nurses and practical nurses).

The aim is to recruit 50 participants, in order to reach a sample of 40 participants in total considering a potential loss to follow-up of 15%.

Educational activities:

The content of the educational activity focuses on maintaining technical skills in positive pressure ventilation (PPV) during neonatal resuscitation and will be based on the contents of the chapter "Positive pressure ventilation" of the "Neonatal resuscitation manual, 8th edition". This activity consists of putting into practice the actions leading to the VPP sequence, as described in the road map, using the T-piece resuscitation machine (Neopuff) and the self-inflating bag, both of which are available in the clinic. It will take place on a mobile training station equipped with the necessary equipment for VPP. Each session will last 30 minutes and will be held during the participants' work shift, thus benefiting from protected time for training, and will be repeated three times over a three-month period.

The teaching strategy varies between the two groups of participants, which are:

1. Intervention group: This approach involves repeated peer-guided practice. Each session will involve two participants, who will support each other using the feedback grid from the first section of the "Neonatal Mask Ventilation Competency Assessment Tool" developed to provide feedback on practising technical skills.
2. Control group: In this group, practice is deliberate (PD) and is led by an instructor. Each session will be supervised by an instructor for two to four participants, and the latter will use the same feedback grid as that used in the intervention group to provide feedback.

Demographic and professional questionnaire:

Following consent to participate in the project, participants will have to complete this questionnaire including demographic data, including age by interval and gender, as well as professional data including work shift (day, evening, night, day and night rotation), initial training (college, university, other), the number of months of experience in neonatology, the approximate number of neonatal resuscitations and positive pressure ventilation in which they participated, the approximate number of simulations in neonatal intensive care in which they participated. These data will be used to describe the characteristics of the study sample.

Performance test (before and after training):

To assess changes in technical skills following the intervention, each participant will be assessed before and after the training.

The assessment will be carried out in the simulation room in the neonatal unit and will last 5 minutes. Upon arrival, the participant will be presented with a clinical vignette of a patient requiring positive pressure ventilation (see appendix). This vignette was created by the project researchers based on their experience in the field of neonatology. After two minutes of positive pressure ventilation, the patient will be stabilized and the vignette will end. A short feedback will be provided to the participant after the evaluation.

Two evaluators, including possibly the researcher himself, will complete the evaluation of each video recording, being blind to the participant's group as well as the phase of the study (pre or post training), using the tool "Neonatal Mask Ventilation Competency Assessment Tool". The effectiveness and relevance of this tool in the evaluation of essential clinical skills has been demonstrated, thus justifying its adoption for the project.

Final questionnaire:

This questionnaire will be completed by the participants at the end of their last practical session and is made up of a first part dedicated to the Continuing Professional Development (CPD) questionnaire and a second which assesses the degree of satisfaction, confidence and feasibility of the tool educational. This data will allow evaluation of th feasibility component, confidence as well as the propensity to change one's practice following th intervention.

ELIGIBILITY:
Inclusion Criteria:

* Registered or practical nurse working in neonatal intensive care at CHU Sainte-Justine
* At least one year of experience in neonatology care at CHU Sainte-Justine
* Completed the initial neonatal resuscitation training

Exclusion Criteria:

* Neonatal transport nurses, due to their particular expertise which may introduce bias.
* Nurse that are instructor for neonatal resuscitation training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction with the quality of the educational methods assessed by a questionnaire | 6 months
  The questionnaire uses a 1 to 4 likert scale with 1 being the highest satisfaction.
Number of participants that agree to participate | 6 months
  From 0 to 50, 50 being the better outcome
Number of participants that terminate the study (retention rate). | 6 months
  From 0 to 50, 50 being the better outcome

SECONDARY OUTCOMES:
Mean difference in performance of VPP as per the Neonatal Mask Ventilation Competency Assessment Tool (NMVCAT) score | 6 months
  Scale from 0 to 100%, higher means better outcome (performance)
Mean difference in confidence level of participants | 6 months
  Likert scale 1 to 4 with 1 being the highest level of confidence
Propensity to change behaviour score based on the CPD-REACTION questionnaire | 6 months
  Rating from 1 to 7, 7 being the highest propensity to change behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Moussa, MD, MMEd, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Dept Neonatology, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No